CLINICAL TRIAL: NCT04567147
Title: Effect of Probiotic on Depressive Symptom in Chinese Patients
Brief Title: Effect of Probiotic on Depression
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: China Agricultural University (Other)
Responsible Party: Principal Investigator, Fazheng Ren, professor, China Agricultural University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAUDepression-01
Record Dates: First submitted 2020-09-20; First posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): Formula probiotic contains freeze-dried Lactobacillus casei, Bafidobacterium animals, Bifidobacterium longum, Bifidobacterium bidium and Lactobacillus plantarum, each at a dosage of 3.0E+10 CFU per 2g sachet.
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo made with only the excipients. The placebo sachet was matched to the study probiotic products for taste, color, and size.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Patients received the formula probiotic for consecutive 8 weeks ( one sachet per day ).
  Arms: Probiotic
Dietary Supplement: Placebo — Patients received the placebo identical to probiotic for consecutive 8 weeks ( one sachet per day ).
  Arms: Placebo

SUMMARY:
Depressive disorder, also known as depression, is a type of mood disorder characterized by persistent low mood. The incidence of depression worldwide is about 6%. Growing evidence suggested that the gut microbiota plays a key role in the development of depression. Probiotics can effectively regulate gut microbiota, and showed potential in alleviating depression. This study investigated the effect of formula probiotic (containing Lactobacillus paracasei, Bifidobacterium animalis, Bifidobacterium longum, Bifidobacterium bifidum and Lactobacillus plantarum) on depression.

ELIGIBILITY:
Inclusion Criteria:

* Normal body mass index ≥ 18.5 until ≤ 29.9
* Mild to moderate major depression diagnosed by psychiatrists according to the diagnostic criteria for depressive episodes in DSM-5 (American Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition))
* Hamilton Rating Scale for Depression (HAMD-17) score not less than 8
* Agreed to intake study product during the study period
* Agreed to sign written informed consent

Exclusion Criteria:

* Use of systemic antibiotics or antimycotics medication in the 30 days prior to the study
* Investigator's uncertainty about the willingness or ability of subject to comply with the protocol requirements
* Persons with a milk protein allergy, lactose intolerance
* Pregnant or breastfeeding women
* Subject had other serious diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-06-22 (Actual); Study Completion 2020-09-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Rating Scale | Changes in the HAMD score at baseline and 8-week intervention
  Depressive symptoms as measured with the Hamilton Rating Scale for Depression. The score rangs from 0 to 53. The higher score means severer depressive symptoms.

SECONDARY OUTCOMES:
Fecal microbiome | Changes between at baseline and 8-week intervention
  changes in the profile of gut microbiota before and after 8-week intervention.
Serum Il-1β | change from baseline to intervention measurements at 8 weeks
  Serum Il-1β levels before and after intervention assessed by ELISA.
Serum Il-6 | change from baseline to intervention measurements at 8 weeks
  Serum Il-6 levels before and after intervention assessed by ELISA.
Serum TNF-α | change from baseline to intervention measurements at 8 weeks
  Serum TNF-α levels before and after intervention assessed by ELISA.
Serum cortisol | change from baseline to intervention measurements at 8 weeks
  Serum cortisol levels before and after intervention assessed by ELISA.
Serum Brain-derived neurotrophic factor | change from baseline to intervention measurements at 8 weeks
  Serum Brain-derived neurotrophic factor levels before and after intervention assessed by ELISA.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Chinese Medicine Hospital Pinggu Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bromet E, Andrade LH, Hwang I, Sampson NA, Alonso J, de Girolamo G, de Graaf R, Demyttenaere K, Hu C, Iwata N, Karam AN, Kaur J, Kostyuchenko S, Lepine JP, Levinson D, Matschinger H, Mora ME, Browne MO, Posada-Villa J, Viana MC, Williams DR, Kessler RC. Cross-national epidemiology of DSM-IV major depressive episode. BMC Med. 2011 Jul 26;9:90. doi: 10.1186/1741-7015-9-90. PMID 21791035
- [Result] Aizawa E, Tsuji H, Asahara T, Takahashi T, Teraishi T, Yoshida S, Ota M, Koga N, Hattori K, Kunugi H. Possible association of Bifidobacterium and Lactobacillus in the gut microbiota of patients with major depressive disorder. J Affect Disord. 2016 Sep 15;202:254-7. doi: 10.1016/j.jad.2016.05.038. Epub 2016 May 24. PMID 27288567
- [Result] Wallace CJK, Milev R. The effects of probiotics on depressive symptoms in humans: a systematic review. Ann Gen Psychiatry. 2017 Feb 20;16:14. doi: 10.1186/s12991-017-0138-2. eCollection 2017. PMID 28239408
- [Result] Kazemi A, Noorbala AA, Azam K, Eskandari MH, Djafarian K. Effect of probiotic and prebiotic vs placebo on psychological outcomes in patients with major depressive disorder: A randomized clinical trial. Clin Nutr. 2019 Apr;38(2):522-528. doi: 10.1016/j.clnu.2018.04.010. Epub 2018 Apr 24. PMID 29731182
- [Result] Akkasheh G, Kashani-Poor Z, Tajabadi-Ebrahimi M, Jafari P, Akbari H, Taghizadeh M, Memarzadeh MR, Asemi Z, Esmaillzadeh A. Clinical and metabolic response to probiotic administration in patients with major depressive disorder: A randomized, double-blind, placebo-controlled trial. Nutrition. 2016 Mar;32(3):315-20. doi: 10.1016/j.nut.2015.09.003. Epub 2015 Sep 28. PMID 26706022